CLINICAL TRIAL: NCT04331496
Title: Saline Serum Versus Hypertonic Serum With Respiratory Physiotherapy in a Recurrent Wheezing Patient: a Multicenter Clinical Trial
Brief Title: Saline vs Hypertonic Serum With Respiratory Physiotherapy in a Recurrent Wheezing Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guadarrama Hospital (Other)
Collaborators: Fisiobronquial Clínicas (Other)
Responsible Party: Principal Investigator, J. Nicolas Cuenca Zaldivar, Rehabilitation Service Principal Investigator, Guadarrama Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8.0
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Bronchiolitis
Keywords: Physical Therapy; Respiratory; Pediatric
MeSH Terms: conditions — Bronchiolitis | interventions — Hypertonic Solutions

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertonic solution (Experimental): Hypertonic solution 4 ml 3% , for 8 minutes in a Philips® vibrating mesh nebulizer plus 20 minute session of Respiratory Physiotherapy based on slow expiratory flow.
  Interventions: Other: Hypertonic solution
- Physiological solution (Active Comparator): Single-dose physiological saline serum (5 ml 0.9% NaCl), for 8 minutes in a Philips® vibrating mesh nebulizer plus 20 minute session of Respiratory Physiotherapy based on slow expiratory flow.
  Interventions: Other: Physiological solution

INTERVENTIONS:
Other: Hypertonic solution — Hypertonic serum 4 ml 3%, administered for 8 minutes in a Philips® vibrating mesh nebulizer plus 20 minute session of Respiratory Physiotherapy based on slow expiratory flow: passive technique of expiratory aid applied to the participant by means of a slow thoracic-abdominal pressure that begins at the end of a spontaneous expiration and continues until the residual volume. The physiotherapist through assisted cough or stimulation of the trachea achieves expectoration of sputum.
  Arms: Hypertonic solution
Other: Physiological solution — Single-dose physiological saline serum (5 ml 0.9% NaCl), administered for 8 minutes in a Philips® vibrating mesh nebulizer plus 20 minute session of Respiratory Physiotherapy based on slow expiratory flow: passive technique of expiratory aid applied to the participant by means of a slow thoracic-abdominal pressure that begins at the end of a spontaneous expiration and continues until the residual volume. The physiotherapist through assisted cough or stimulation of the trachea achieves expectoration of sputum.
  Arms: Physiological solution

SUMMARY:
Bronchiolitis (BQ) is an acute viral infection of the lower respiratory tract that affects the bronchioles of babies younger than 24 months of age. Respiratory physiotherapy (FTR) appears as a complementary treatment measure in clinical guidelines and consensus on the management of BQ. Nebulization with 3% hypertonic serum before the FTR session induces an osmotic flow of water in the mucus, which facilitates drainage and reduces edema in the submucosal tissue.

DETAILED DESCRIPTION:
Once each patient legal guardians has signed the informed consent document and it has been verified that the inclusion criteria are met, participants will be assigned the same identification number (ID) that is related to its Clinical History (CH) by simple coding; custody of the file with the relationship of each ID with its CH will be the responsibility of the principal investigator. The method of blinding in the allocation will be carried out by choosing envelopes sealed by an external investigator to the study. The contents of the envelopes will be randomized by computer using the numerical randomization sequence generated with R ver 5.3.1 (R Foundation for Statistical Computing, Institute for Statistics and Mathematics, Welthandelsplatz 1, 1020 Vienna, Austria) based on stratified sampling for homogeneity , in two groups: nebulization with 3% hypertonic solution (group A) and in the nebulization group with 0.9% saline solution (group B).

None of the participants who make up both the control and intervention groups will be prohibited from regular pharmacological treatment as prescribed by their doctor, such as Ventolin. It will be collected in the investigator's notebook the medications that each patient has prescribed by their doctor. But applying a bronchodilator is not part of the protocol, because physiotherapists cannot prescribe or administer a drug. Before receiving the usual and standard manual techniques of respiratory physiotherapy, patients receive nebulization, group A with hypertonic serum 4 ml 3% and group B with a single-dose saline (0.9 NaCl) physiological serum 5 ml for 8 minutes, both with nebulizer Philips® vibrating mesh. The effects of both are similar in effects, in terms of secretions and their osmotic effects. The aim of this study is to evaluate if the type of serum affects the results of the manual physiotherapy that is later carried out on children, but there is no clinical problem for randomly giving one serum or another, as to what is the effect of the serum on itself.

The intervention ends with a 20-minute session of Respiratory Physiotherapy based on slow expiratory flow: a passive technique of expiratory aid applied to the participants by means of slow thoracic-abdominal pressure that begins at the end of a spontaneous expiration and continues until the residual volume. The physiotherapist through assisted cough or stimulation of the trachea achieves expectoration of sputum. Care must be taken during the maneuvers to maintain a supine position of the patient in a 30-degree incline, to avoid episodes of gastroesophageal reflux and decrease the risk of vomiting.

Both groups will receive 3 evaluations by an investigator who will be blinded on the treatment and the objectives. The evaluations will be carried out at the beginning of the session (T0), immediately after the nebulization (T30) and 10 minutes after the end of the 20-minute physical therapy intervention (T60). This same treatment and evaluation sequence will be carried out every month for 6 months.

The main variables will classify the participants according to the initial clinical severity score proposed by Wang (WS), the Wood-Downes Scale modified by Ferres (WDF-S) and the Pulmonary Score (PS) in addition to the measurement of Sp2 and heart rate (FC) measured through a pulse oximeter (Radical Touchscreen from Massimo®, Masimo Corporation, Irvine, CA)

ELIGIBILITY:
Inclusion Criteria:

* Have a medical diagnosis of a recurrent wheezing.
* Have the informed consent signed by the legal guardians of the kid.

Exclusion Criteria:

* Acute bronchitis with score> 9 according to the Wang and Pulmonary Score clinical scale.
* Acute BQ with score> 8 on Ferres' modified Wood-Downes scale (WDF-S)
* Parental refusal
* Comorbidity as cardiac, neurological or traumatic pathology.
* Congenital anomalies.
* Chronic pulmonary pathology such as bronchodysplasia.
* Severe obstruction with a punctuation >10 according ESBA and >7 according pulmonary score.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-04-04 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Modified Wang clinical severity scale | 6 months
  The clinical severity scale of Wang evaluates the respiratory rate, the presence of wheezing and intercostal retraction, and the patient's general condition, puncturing each dimension from 0 (the possible state) to 3 (values within normal), in addition to offer different cut points for children with more or less than 6 months.

SECONDARY OUTCOMES:
Pulmonary Score | 6 months
  It is a scale that is used to assess the severity of asthmatic exacerbation in children. The clinical severity scoring system is made up of three items: FR (by age), wheezing, and use of accessory musculature (sternocleidomastoid). Each item is scored from 0 to 3, the values of each item are added and a total result is obtained that goes from 0 (without exacerbation or very slight) to 9 (severe exacerbation).
Wood-Downes scale modified by Ferres | 6 months
  Is a quantitative cumulative scale designed to assess clinical severity in patients with BQ. The clinical severity scoring system consists of six items: wheezing, circulation, respiratory rate (RF), heart rate (HR), ventilation, and cyanosis. Each item is scored from 0 to 3, the values of each item are added together and a total result of (1-3) mild, (4-7) moderate and (> 8) severe is obtained, with 14 being the maximum score and 0 the minimum. A higher score indicates a worse condition.
Oxygen saturation | 6 months
  Measured by a pulse oximeter (Radical 7 Touchscreen by Massimo®, Masimo Corporation, Irvine, CA).
Heart rate | 6 months
  Measured by a pulse oximeter (Radical 7 Touchscreen by Massimo®, Masimo Corporation, Irvine, CA).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Nicolas Cuenca Zaldivar, Mr, Principal Investigator — Hospital Guadarrama, servicio de fisioterapia
Locations (1):
- J.Nicolas Cuenca Zaldivar, Guadarrama, Madrid, Spain

REFERENCES:
- [Derived] Gonzalez-Bellido V, Velaz-Baza V, Rama-Suarez N, Jimeno-Esteo C, Sirvent-Gomez J, Cuenca-Zaldivar JN, Mayorales-Lises S, Donadio MVF, Fernandez-Carnero S. Effects and safety of hypertonic saline combined with airway clearance in non-hospitalized children with recurrent wheezing. Hong Kong Physiother J. 2023 Dec;43(2):105-115. doi: 10.1142/S1013702523500105. Epub 2023 Apr 14. PMID 37583920